CLINICAL TRIAL: NCT05040815
Title: A Prospective Phase II Study of Inguinal Node Sparing Radiotherapy For Patients With Early Stage Anal Cancer (INSPIRE)
Brief Title: Inguinal Node Sparing Radiotherapy For Patients With Early Stage Anal Cancer
Acronym: INSPIRE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-0021
Record Dates: First submitted 2021-06-29; First posted 2021-09-10 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Anal Canal Cancer
Keywords: radiotherapy
MeSH Terms: conditions — Anal Canal Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- chemo-radiation treatment (Experimental): Radiotherapy with concurrent 5-fluorouracil and mitomycin-C combination treatment.
  Radiotherapy consists of 5400 cGy delivered in 30 fractions over 6 weeks. The investigators will be using the current standard regimen for the study or no change in the current CCI treatment regimen. However, the radiotherapy target will be smaller than current practice since the investigators will be omitting prophylactic inguinal irradiation.
  Interventions: Radiation: chemo-radiation treatment

INTERVENTIONS:
Radiation: chemo-radiation treatment — Radiotherapy (RT) with concurrent 5-fluorouracil and mitomycin-C (5FU/MMC) combination is the treatment of choice for non-metastatic locally advanced anal squam

SUMMARY:
The purpose of this study is to see whether avoiding preventative radiation to the groin in patients with normal sentinel node biopsy and PET-CT, is at least as effective treating cancer as giving preventative radiation to the groin for patients with anal canal cancer.

The investigators also want to know if avoiding radiation to the groin will cause fewer side effects and better quality of life

DETAILED DESCRIPTION:
Radiotherapy (RT) with concurrent 5-fluorouracil and mitomycin-C (5FU/MMC) combination is the treatment of choice for non-metastatic locally advanced anal squamous cell carcinoma (ASCC). While, locally advanced AC treatment involves elective inguinal lymph node irradiation along with concurrent chemotherapy with significant improvement of locoregional control and colostomy free survival, many oncologists believe that routine, elective irradiation of bilateral inguinal areas of patients with limited disease (T1-T3) without lymph node involvement may be overtreatment and the larger radiation target that includes entire pelvis and bilateral inguinal region causes significant acute and late toxicities.

SLNB is the standard procedure currently used for breast cancer staging. The most significant observation was that when the SLN is negative, no further ALND or adjuvant axillary radiation is need for those patients. The SLNB had shown a better diagnostic accuracy (31% vs.25%) and higher sensitivity (85% vs.75%) than FDG-PET imaging to detect inguinal lymph node metastasis. Given better diagnostic accuracy and high sensitivity of SLNB, this technique could be used precisely to define target population who could be spared of prophylactic inguinal irradiation.

The investigators hypothesize that patients with early clinical stage node negative anal cancer (T1-T3N0) have low risk of subclinical inguinal lymph node involvement that can be detected by a combination of PET imaging and SLNB. Hence, any early stage AC patients with node negative disease confirmed by PET imaging and SLNB have relatively low risk of nodal failure and so inguinal radiation could be avoided. This approach would limit over treatment of early stage patients, reduce acute and late toxicities. This will be tested in a phase II study with close follow up of study patients so that inguinal relapse if any occur will be salvaged successfully. If this treatment approach is successful, it could be practice changing with improvement of H-QOL of patient.

ELIGIBILITY:
Inclusion Criteria:

1. Participants capable of giving informed consent.
2. Patients must be 18 years of age or older.
3. Patient should have histologically proven primary squamous cell carcinoma.
4. Patients must have early AC, Stage T1-3 N0 M0.
5. No inguinal nodal involvement confirmed by PET imaging and SLNB.
6. No history of prior malignancy other than non-melanoma skin cancer or other malignancy with disease free survival ≥ 5 years.
7. Performance status ECOG 0-2 / Zubrod performance status ≥70.
8. Patient should be eligible for concomitant chemotherapy (e.g. adequate hepatic, renal and bone marrow function).
9. Women of child bearing potential (WOCBP) must have a negative serum (or urine) pregnancy test at the time of screening. WOCBP is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy or bilateral salpingectomy) and is not postmenopausal. Menopause is defined as 12 months of amenorrhea in a woman over age 45 years in the absence of other biological or physiological causes. In addition, females under the age of 55 years must have a serum follicle stimulating hormone, (FSH) level > 40 mIU/mL to confirm menopause.
10. Patients of childbearing / reproductive potential should use highly effective birth control methods, as defined by the investigator, during the study treatment period. A highly effective method of birth control is defined as those that result in low failure rate (i.e. less than 1% per year) when used consistently and correctly (Note: abstinence is acceptable if this is established and preferred contraception for the patient and is accepted as a local standard).
11. Females must not breastfeed during study treatment.
12. Male patients should agree to not donate sperm during study treatment.
13. Absence of any condition hampering compliance with study protocols and follow-up schedule; those conditions should be reviewed with the patient prior to trial registration.

Exclusion Criteria:

1. T1N0 patients going for primary surgery
2. Prior radiation therapy to the pelvis.
3. Pregnancy or lactation.
4. Prior surgical treatment for anal cancer other than biopsy.
5. Prior surgical or chemotherapy treatment for anal cancer.
6. Evidence of distant metastases.
7. Comorbid medical conditions precluding radical treatment at the discretion of Oncologist.
8. Histology other than squamous cell carcinoma or variants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-05-11 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of inguinal lymph node recurrence | Total duration of follow up is 36 months
  The primary end point is measured by PET/CT imaging at 3 months post treatment and, then CT scan of chest, abdomen and pelvis every 3 months for 2 years and then every 6 months for another year.
Disease free survival (DFS) | 36 months
  Time between enrollment and date of relapse (radiographic or clinical progression) leading to change in therapy for recurrent disease or death due to any cause.

SECONDARY OUTCOMES:
Health related Quality of Life (EORTC QLQ-C30) | 36 months
  Evaluation will be done using EORTC QLQ-C30 (European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire C30). Assessed at baseline (before starting CRT) and, at 3 months, 12 months, 24 months and 36 months after completion of treatment.
Health related Quality of Life (EORTC QLQ-AN27) | 36 months
  Evaluation will be done using EORTC QLQ-AN27, the supplementary module specific for anal cancer. Assessed at baseline (before starting CRT) and, at 3 months, 12 months, 24 months and 36 months after completion of treatment.
Health related Quality of Life (IIEF) | 36 months
  Evaluation will be done using International Index of Erectile Function (IIEF) for Men. Assessed at baseline (before starting CRT) and, at 3 months, 12 months, 24 months and 36 months after completion of treatment.
Health related Quality of Life (FSFI) | 36 months
  Evaluation will be done using Female Sexual Function Index (FSFI). Assessed at baseline (before starting CRT) and, at 3 months, 12 months, 24 months and 36 months after completion of treatment.
Health related Quality of Life (Vaizey Score) | 36 months
  Evaluation will be done using Vaizey Score to analyse severity of anal incontinence. Assessed at baseline (before starting CRT) and, at 3 months, 12 months, 24 months and 36 months after completion of treatment.
Health related Quality of Life (Fecal Incontinence Severity Index) | 36 months
  Evaluation will be done using Fecal Incontinence Severity Index. Assessed at baseline (before starting CRT) and, at 3 months, 12 months, 24 months and 36 months after completion of treatment.
Treatment-related acute toxicities | Up to 3 months
  Treatment-related acute toxicity will be assessed based on the acute morbidity criteria by NCI CTCAE v.5.0. Acute treatment related morbidity will be assessed weekly during treatment. Then 3 months after completion of treatment.
Treatment-related late toxicities. | 36 months
  Late morbidity is defined as morbidity occurring 90 days after completion of treatment. Treatment-related late toxicities will be assessed every 3 months for 2 years and every 6 months for another year.
Exercise Behavior and Physical Fitness | 36 months
  Self-reported exercise behavior will be measured before treatment, after treatment, and at 4 months, 8 months, 1-year, 2-year, and 3-year follow-up using the Godin Leisure-Time Exercise Questionnaire [36]. Objective physical fitness will be measured before treatment, after treatment, and at 4 months and 1-year follow-up using the Senior's Fitness Test (SFT) [37, 38]. The SFT consists of: (a) 30-second chair stand, (b) 30-second arm curl, (c) chair sit-and-reach, (d) back scratch, (e) 8-foot up-and-go, and (f) 6-minute walk. These tests, respectively, assess lower and upper body strength, lower and upper body flexibility, agility/dynamic balance, and aerobic endurance.

OTHER OUTCOMES:
Relationship between radiotherapy treatment planning variables and acute toxicity. | 36 months
  We will be collecting information related to treatment plans for each patient such as total irradiated volume, dose to OARs, integral dose and will evaluate any association between these factors and toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Kurian Joseph, MD, Principal Investigator — AHS-CCI
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada